CLINICAL TRIAL: NCT02634021
Title: Hemodynamic Change Between Loading of Dexmedetomidine or Midazolam as a Sedative Agents During Knee Arthroscopy
Brief Title: Effect of Loading of Midazolam or Dexmedetomidine on Hemodynamics
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The investigator had no more scientific interest about this issue.
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Seong-Hyop Kim, Professor, Konkuk University Medical Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: KUH1160088
Record Dates: First submitted 2015-12-09; First posted 2015-12-17 (Estimated); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Knee Injuries
MeSH Terms: conditions — Knee Injuries | interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexmedetomidine group (Active Comparator): dexmedetomidine 1 mcg/kg intravenous loading followed by dexmedetomidine continuous infusion at the rate of 0.5 mcg/kg/hr
  Interventions: Drug: dexmedetomidine group
- midazolam group (Experimental): midazolam 0.1 mg/kg intravenous loading followed by dexmedetomidine continuous infusion at the rate of 0.5 mcg/kg/hr
  Interventions: Drug: midazolam group

INTERVENTIONS:
Drug: dexmedetomidine group — intravenous loading of dexmedetomidine for 1 mcg/kg
  Other Names: dexmedetomidine
  Arms: dexmedetomidine group
Drug: midazolam group — intravenous loading of midazolam for 0.1 mg/kg
  Other Names: midazolam
  Arms: midazolam group

SUMMARY:
Loading dose of dexmedetomidine is related hemodynamic instability such as bradycardia and hypertension.

DETAILED DESCRIPTION:
The investigators hypothesized substitution of loading of dexmedetomidine for midazolam could reduce hemodynamic instability during spinal anesthesia for knee arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

* patients who were planned to undergo knee arthroscopy under spinal anesthesia

Exclusion Criteria:

* age < 20 years
* underlying heart, liver or kidney disease
* hypersensitivity to midazolam or dexmedetomidine

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
change of heart rate | from 1 minute before anesthesia to 1 hr after anesthesia

SECONDARY OUTCOMES:
change of bispectral index | from 1 minute before anesthesia to 1 hr after anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Seong-Hyop Kim, Professor, Principal Investigator — Konkuk University Medical Center
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No